CLINICAL TRIAL: NCT06148129
Title: Stratification of Endometrial Carcinoma Patients Using Immunohistochemistry for Better Surgical Planning and Prognosis
Brief Title: Immunohistochemistry Role in Better Prognosis of Endometrial Carcinoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Walid Mohamed Elnagar, Assistant professor of gynecology, Zagazig University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB#10903-21/6-2023
Record Dates: First submitted 2023-11-13; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator)
  Interventions: Diagnostic Test: Tissue Biopsy
- Excluded Patients (No Intervention)

INTERVENTIONS:
Diagnostic Test: Tissue Biopsy — The Post-hysterectomy tissue biopsy was analyzed immunohistochemically for detection of estrogen and progesterone receptors, P53 and L1CAM
  Arms: Study group

SUMMARY:
The incidence of endometrial cancer (EC) is increasing .Different risk classifications are used to direct the primary and adjuvant therapy. The European Society for Medical Oncology - European Society of Gynaecological Oncology -European Society for Radiotherapy & Oncology (ESMO-ESGO- ESTRO) could guide the need for lymph node surgery pre-operatively, and also post-operatively to determine adjuvant treatment.

Low-risk patients are managed with surgery alone, while higher-risk group patients undergo more aggressive surgical options. So, it is important to identify new prognostic markers for better stratification of patients to avoid under- or over treatment of EC patients.

ELIGIBILITY:
Inclusion Criteria:

* aged 36 -72 years;
* Previously diagnosed with endometrial carcinoma;
* Histological Type of the tumor;
* Myometrial Invasion;
* lymph Node Invasion;
* Cervical Invasion;
* Biomarkers expression.

Exclusion Criteria:

* Lack of tumor tissue in tissue block

Ages: 36 Years to 72 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
expression levels of p53/L1CAM/ER/PR | 36 Months
  The Prognostic value of immunohistochemical detection of expression levels of p53/L1CAM/ER/PR in relation to ESMO-ESGO-ESTRO risk groups

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university, Zagazig, Ash Sharqia Governorate, Egypt